CLINICAL TRIAL: NCT04884061
Title: Description of the Vasculature Pattern of the Bronchial Tree During Infection With SARS-CoV2 by Narrow Band Imaging Bronchoscopy
Brief Title: Narrow Band Imaging Bronchoscopy During SARS-CoV2 Infection
Acronym: SARS-CoV2-NBI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0096
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Covid19; Bronchoscopy; Narrow-band Imaging
Keywords: Covid19; bronchoscopy; Narrow-band imaging; bronchial vasculature; Acute vascular distress syndrome
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental: Patients hospitalized with SARS-CoV2 infection proven by RT-PCR test
  Interventions: Other: NBI images and/or videos
- Comparator: Patients hospitalized with lower respiratory tract infections unrelated to SARS-CoV2 (RT-PCR negative for SARS-CoV2)
  Interventions: Other: NBI images and/or videos
- Comparator 2: Patients who have had bronchoscopy performed as part of the assessment of a distal pulmonary nodule (RT-PCR negative for SARS-CoV2).
  Interventions: Other: NBI images and/or videos

INTERVENTIONS:
Other: NBI images and/or videos — A library of NBI images and/or videos will be established from previously recorded bronchoscopies in 30 patients (10 with a SARS-CoV2 infection, 10 with a lower respiratory tract infection not related to SARS-CoV2, and 10 in patients with pulmonary nodule). NBI images and/or videos of the bronchial tree will then be analysed by three experimented interventional pulmonologists blinded to the patient ID. Each investigator will describe the vasculature pattern according to a prespecified grid: Normal mucosal vascularity / increased capillary density / presence of capillary loops / presence of dotted vessels / complex vascular networks of tortuous vessels or abrupt ending vessels / dilated longitudinal vessels. In case of discordance between the investigators, images will be reviewed to obtain a consensus.

SUMMARY:
Vascular modifications have been described during SARS-CoV2 infection, especially a dilatation of the bronchial arteries. Within the airway wall, small branches of the bronchial arteries cross the muscle layer to develop a submucosal network. The Narrow Band Imaging technique is used during bronchoscopy to achieve a maximum contrast of vessels and the surrounding mucosa. Therefore, it enables to observe the microvessel structure and its distribution in the bronchial mucosa. The aim of this study is to describe the vasculature pattern of the bronchial tree during infection with SARS-CoV2.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo bronchoscopy with image and/or videos recording of NBI aspect of the proximal bronchial tree (carina, right and left upper lobe).
* Patients hospitalized with SARS-CoV2 infection proven by RT-PCR test
* patients hospitalized with lower respiratory tract infections unrelated to SARS-CoV2 (RT-PCR negative for SARS-CoV2)
* Patients who have had bronchoscopy performed as part of the assessment of a distal pulmonary nodule (RT-PCR negative for SARS-CoV2).

Exclusion Criteria:

* Patients under legal protection
* Patients who refuses the use of his personal medical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients who undergo bronchoscopy with image and/or videos recording of NBI aspect of the proximal bronchial tree (carina, right and left upper lobe). Three groups of patients will be selected: 1) Patients hospitalized with SARS-CoV2 infection proven by RT-PCR test ; 2) patients hospitalized with lower respiratory tract infections unrelated to SARS-CoV2 (RT-PCR negative for SARS-CoV2) ; 3) Patients who have had bronchoscopy performed as part of the assessment of a distal pulmonary nodule (RT-PCR negative for SARS-CoV2).
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Variation of the vasculature pattern of the bronchial mucosa between the three patient groups | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No